CLINICAL TRIAL: NCT01827137
Title: A Pilot Trial of a WT1 Analog Peptide Vaccine in Patients With Multiple Myeloma Following Autologous Stem Cell Transplantation
Brief Title: WT1 Vaccine Treatment of Patients With Multiple Myeloma After Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sellas Life Sciences Group (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-288
Expanded Access: NCT05593185 (Available)
Record Dates: First submitted 2013-04-02; First posted 2013-04-09 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple Myeloma
Keywords: WT1 Analog Peptide Vaccine; 12-288; Galinpepimut-S; GPS; Maintenance therapy; Autologous Stem Cell Transplant (ASCT); Wilms Tumor 1; Immunotherapeutic Agent; Post-ASCT maintenance; SLS-001
MeSH Terms: conditions — Multiple Myeloma; Wilms Tumor | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Monatide (IMS 3015); Lenalidomide; Immunomodulating Agents; Bortezomib; Proteasome Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Galinpepimut-S + Montanide + GM-CSF (Experimental): Galinpepimut-S (GPS) vaccinations are started 12-22 days following autologous stem cell transplantation (ASCT). GPS and Montanide (in a 1 mL emulsion) are administered subcutaneously (s.c.) Q2W on weeks 0, 2, 4, 6, 8, and 10. GM-CSF (70 μg) are administered s.c. one to two days before and on the day of GPS/Montanide administration. Participants whose disease has not progressed and who are clinically stable (no active infection with fevers and no cardiovascular/respiratory compromise) may receive up to 6 additional monthly vaccinations. The use of post-ASCT maintenance therapy is allowed starting 3 months after ASCT.
  Interventions: Biological: Galinpepimut-S; Biological: GM-CSF; Other: Montanide; Drug: lenalidomide; Drug: bortezomib

INTERVENTIONS:
Biological: Galinpepimut-S — Galinpepimut-S admixed with the adjuvant Montanide following specified schedule
  Other Names: GPS; SLS-001
Biological: GM-CSF — subcutaneous injection
  Other Names: sargramostim
Other: Montanide — adjuvant
Drug: lenalidomide — optional post-ASCT therapy
  Other Names: immunomodulatory drugs
Drug: bortezomib — optional post-ASCT therapy
  Other Names: proteasome inhibitor

SUMMARY:
The purpose of this trial is to assess the immune response after vaccination with a peptide vaccine called galinpepimut-S (or GPS) in a type of blood cancer called multiple myeloma. A protein called WT1 is often present in cancerous cells and GPS can train the immune system to recognize and kill the cancerous cells containing WT1. This study will also assess the safety of GPS, effect on disease, and on survival.

Participants who has undergone autologous stem cell transplant (ASCT) will receive vaccinations with GPS every 2 weeks for 10 weeks (a total of 6 vaccinations). Vaccinations will start 12 to 22 days after ASCT. In the absence of disease progression and if clinically stable after the first 6 vaccinations, participants may continue to receive six more vaccinations every month. The use of post-ASCT maintenance therapy is allowed starting from 3 months after transplant.

DETAILED DESCRIPTION:
This is an early phase clinical study conducted in patients with newly diagnosed high-risk multiple myeloma to examine the effects of vaccination with galinpepimut-S (GPS) on clinical and immunobiological indices. The study is titled "A Pilot Trial of a WT1 Analog Peptide Vaccine (Galinpepimut-S) in Patients With Multiple Myeloma Following Autologous Stem Cell Transplantation" and is designed as a single-arm, single-institution, open-label study. The primary objective is to assess immune response 12 to 14 weeks after administration of GPS in patients with new diagnosed multiple myeloma (MM) following autologous stem cell transplant (ASCT). Secondary objective includes assessing the safety profile, progression-free survival, and overall survival.

Galinpepimut-S (GPS) consists of four WT1-derived peptides which have been chosen to strengthen antigenicity, but also broaden immunogenicity over a wide range of HLA subtypes, being able to stimulate both CD8+ (MHC Class I)- and CD4+ (MHC Class II)-dependent responses. Galinpepimut-S is administered with the adjuvant Montanide and sargramostim (GM-CSF).

Participants who has undergone autologous stem cell transplant (ASCT) will receive vaccinations with GPS every 2 weeks for 10 weeks (a total of 6 vaccinations). Vaccinations will start 12 to 22 days after ASCT. In the absence of disease progression and if clinically stable after the first 6 vaccinations, participants may continue to receive six more vaccinations every month. The use of post-ASCT maintenance therapy with immunomodulatory drugs (IMIDs, eg, thalidomide, lenalidomide) or proteasome inhibitors (PSIs, eg, bortezomib) is allowed from 3 months after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma, ISS stage 1-3 with confirmed diagnosis of multiple myeloma at MSKCC
* Patients must be eligible to undergo autologous stem cell transplantation by standard institutional criteria
* Patients must have documented WT1 positive disease. For purpose of this study, this is defined as detectable presence of WT1 expression by immunohistochemistry or by WT1 transcript via RT-PCR on a bone marrow or other plasma cell-related biopsy specimen prior to autologous stem cell transplantation. Bone marrow or other biopsy specimen from time of diagnosis from patients diagnosed at MSKCC or outside hospital may be requested for assessment of WT1 expression by IHC
* Age > or = to 18 years
* Karnofsky performance status > or = to 50%
* Hematologic parameters:
* Absolute neutrophil count (ANC) > or = to 1,000/μl
* Platelets > 50,000/μl
* Biochemical parameters:
* Total bilirubin < than or = to 2.0 mg/dl
* AST and ALT < than or = to 2.5 x upper limits of normal (ULN)
* Creatinine < than or = to 2.0 mg/dl

Exclusion Criteria:

* Pregnant or lactating women
* Patients with active infection requiring systemic antimicrobials
* Patients taking systemic corticosteroids
* Patients with serious unstable medical illness
* Concurrent malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2017-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Koehne, MD, PhD, Study Director — Miami Cancer Institute (Baptist Health South Florida) - formerly at MSKCC; David J Chung, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koehne G, Devlin S, Korde N, Mailankody S, Landau H, Hassoun H, Lesokhin A, Lendvai N, Chung D, Sarlis N, Giralt S, Landgren O. Galinpepimut-S, a WT1-Targeting Immuno-Oncology Treatment, Induces Specific, Robust and Durable Immune Responses (IRs) in Patients (Pts) with High-Risk (HR) Multiple Myeloma (MM). Clinical Lymphoma, Myeloma and Leukemia 17: S343-S344, 2017
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Analysis set
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 61.3 [46 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Type of myeloma [Count of Participants; unit: Participants]
  IgG | 12
  IgA | 4
  Light chain | 3
Prior therapies [Median (Full Range); unit: number of therapies] | 2 [1 to 3]
Post ASCT therapy [Count of Participants; unit: Participants]
  Lenalidomide alone or in combination | 18
  Other (bortezomib) | 1
Prior ASCT [Count of Participants; unit: Participants]
  1 | 17
  2 | 2
Cytogenetics at diagnosis [Count of Participants; unit: Participants]
  High risk | 15
  Average risk | 4

OUTCOME MEASURES:

1. Primary Outcome: WT1 T-cell Immune Response (IR) 12-14 Weeks After First GPS Administration (6 x Administrations)
Description: Number and percentage of participants with CD4 and/or CD8 immune responses against WT1m measured 12-14 weeks after first GPS administration (6 x administrations)
Time Frame: 12 weeks after the initial GPS vaccine (end of first series [GPS x 6 administrations])
Population: Only 15 patients completed 6 x GPS administrations
Measure: Count of Participants; unit: Participants
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Number analyzed (Participants) | 15
Participants | 9

2. Secondary Outcome: Progression-free Survival (PFS) From Autologous Stem Cell Transplant (ASCT)
Description: PFS measured from ASCT to time of myeloma progression (as defined by the International Myeloma Working Group [IMW] consensus criteria or subject death.
Time Frame: 3 years and 8 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Number analyzed (Participants) | 19
days | 717 [286 to NA] — Upper 95%CI not reached due to end of study monitoring duration

3. Secondary Outcome: Overall Survival (OS) From Autologous Stem Cell Transplant (ASCT)
Description: OS measured from time of autologous stem cell transplant (ASCT) to the time of subject death
Time Frame: 3 years and 8 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Number analyzed (Participants) | 19
days | NA [NA to NA] — Median OS and 95% CI not reached due to end of the study monitoring period (3 years and 8 months)

4. Post Hoc Outcome: WT1 T-cell Immune Response (IR) After Completion of All GPS Administrations
Description: Number and percentage of participants with CD4 and/or CD8 immune responses against WT1 measured after all GPS administrations (12 x administrations)
Time Frame: 38 weeks after the initial GPS vaccine (end of booster series [GPS x 12 administrations])
Population: 12 patients completed all 12 x GPS administrations
Measure: Count of Participants; unit: Participants
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: 4.5 years
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Galinpepimut-S + Montanide + GM-CSF (N=20)
Anemia (Blood and lymphatic system disorders) | 20
Hyperglycemia (Metabolism and nutrition disorders) | 20
Hypoalbuminemia (Metabolism and nutrition disorders) | 20
Lymphocyte count decreased (Investigations) | 20
Neutrophil count decreased (Investigations) | 20
Platelet count decreased (Investigations) | 20
White blood cell decreased (Investigations) | 20
Hypocalcemia (Metabolism and nutrition disorders) | 19
Alanine aminotransferase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 12
Hypokalemia (Metabolism and nutrition disorders) | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Fatigue (General disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 9
Alkaline phosphatase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 8
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypernatremia (Metabolism and nutrition disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Cholesterol high (Investigations) | 5
Creatinine increased (Investigations) | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 4
INR increased (Investigations) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Anxiety (Psychiatric disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Nervous system disorders - Other, (Nervous system disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Injection site reaction (General disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes